CLINICAL TRIAL: NCT00919594
Title: Psychotherapy for Depressed Mothers of Psychiatrically Ill
Brief Title: Psychotherapy for Depressed Mothers of Psychiatrically Ill Children
Acronym: IPT-MOMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Holly Swartz, Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO08100448; 5R01MH083647 (NIH)
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Depression
Keywords: Interpersonal Psychotherapy; Depression; Mothers
MeSH Terms: conditions — Depression | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interpersonal Psychotherapy for Mothers (Experimental): Interventions will be administered during the 3 Month Acute Randomized Phase and will consist of nine individual 45-minute sessions conducted over the course of three months. Treatment cannot exceed nine sessions. In addition to standard IPT techniques, IPT-MOMS includes a specific focus on the challenges associated with managing a child who suffers from psychiatric problems.
  Interventions: Behavioral: Interpersonal Psychotherapy for Mothers (IPT-MOMS)
- Brief Supportive Psychotherapy (Active Comparator): Interventions will be administered during the 3 Month Acute Randomized Phase and will consist of nine individual 45-minute sessions conducted over the course of three months. Treatment cannot exceed 9 sessions. Brief supportive therapy (BSP) is a manualized form of supportive psychotherapy which emphasizes reflective listening and elicitation of affect (Markowitz et al., 2008). Therapists are instructed to allow patients to determine the focus of each session, pulling for emotion, validating emotions when possible, and offering empathic comments.
  Interventions: Behavioral: Brief Supportive Psychotherapy

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy for Mothers (IPT-MOMS) — Interventions will be administered during the 3 Month Acute Randomized Phase and will consist of nine individual 45-minute sessions conducted over the course of three months. Treatment cannot exceed nine sessions. In addition to standard IPT techniques, IPT-MOMS includes a specific focus on the challenges associated with managing a child who suffers from psychiatric problems.
  Arms: Interpersonal Psychotherapy for Mothers
Behavioral: Brief Supportive Psychotherapy — Interventions will be administered during the 3 Month Acute Randomized Phase and will consist of nine individual 45-minute sessions conducted over the course of three months. Treatment cannot exceed 9 sessions. Brief supportive therapy (BSP) is a manualized form of supportive psychotherapy which emphasizes reflective listening and elicitation of affect (Markowitz et al., 2008). Therapists are instructed to allow patients to determine the focus of each session, pulling for emotion, validating emotions when possible, and offering empathic comments.
  Arms: Brief Supportive Psychotherapy

SUMMARY:
The current proposal is a randomized, controlled, clinical trial to evaluate the intergenerational impact of treating depressed mothers whose children suffer from psychiatric disorders.

DETAILED DESCRIPTION:
This study will compare a psychotherapy for mothers that targets factors known to be associated with the intergenerational transmission of psychiatric disorders to a nonspecific psychotherapeutic control condition. It will evaluate outcomes in both children and mothers. A modified form of interpersonal psychotherapy for depression, IPT-MOMS, specifically addresses maternal depressive symptoms, maternal interpersonal functioning, and mother-child communication, all factors that contribute to psychiatric illness in youth (Swartz et al., 2006). This application proposes to recruit mother-child dyads, both of whom suffer from psychiatric illness, randomly assign mothers to nine sessions over 3 months of either IPT-MOMS (N=105) or brief supportive psychotherapy (BSP; N=105), and evaluate the impact of acute maternal treatment on child and maternal outcomes at 3, 6, 9, and 12 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria (Mothers)

1. Adult female, age 18-65
2. Biological or adoptive mother of child, age 7-18, who meets child inclusion criteria (see below)
3. Lives with and has custody of the eligible child participant
4. Currently in an episode of major depression, as defined by the DSM-IV and documented by the use of the Structured Clinical Interview for Axis I DSM-IV Disorders (SCID-I)
5. Score > or equal to 15 on the 25-item Hamilton Rating Scale for Depression (HRSD-25)
6. Ability and willingness to give informed, written consent
7. Willingness to give informed consent for their eligible and assenting child to participate

Inclusion Criteria (Psychiatrically Ill Children)

1. Age 7-18
2. Currently meets criteria for at least one current depressive or anxiety disorder as defined by the DSM-IV (American Psychiatric Association, 1994) and documented by the Schedule for Affective Disorders and Schizophrenia for School Age Children, Present and Lifetime version (K-SADS-PL)
3. Willingness to provide informed consent/assent

Exclusion Criteria:

Exclusion Criteria (Mothers)

1. If a mother subject IS NOT on antidepressants:

   Mothers must be off all antidepressant medications for at least 14 days (30 days for fluoxetine) prior to screening to ensure that pretreatment assessments are not distorted by drug withdrawal or rebound effects). Mother subjects cannot start taking antidepressant medications during the acute treatment phase. If they do start taking antidepressant medication during the acute treatment portion of the study, their participation in the acute phase of the study will be terminated. They will be continued to be followed in the follow-up phase.

   If a mother subject IS on antidepressants:

   Mothers must be on a stable dose of an antidepressant medication (4 consecutive weeks at the same dose) prior to signing consent. The mother subject must agree to stay on the same antidepressant at this current dose throughout the duration of the acute phase of the study. If a participant's dosage of an antidepressant medication is changed or if they cease taking their antidepressant medication during the acute treatment portion of the study, their participation in the acute phase of the study will be terminated. They will be continued to be followed in the follow-up phase.
2. Active suicidal ideation or homicidal ideation that in the clinical opinion of the research team as headed by the PI, would require hospitalization
3. At serious risk for child abuse or neglect which in the clinical opinion of the research team as headed by the PI, requires intervention
4. Comorbid psychotic disorder, organic mental disorder, current (within prior six months) substance or alcohol abuse, borderline personality disorder, antisocial personality disorder, or history of a prior manic episode (bipolar disorder)
5. Significant medical illness that might explain depressive symptoms such as epilepsy, autoimmune disorders, or unstable endocrine disease
6. Not fluent in English. The intervention to be tested in this study is psychotherapy. The staff is only trained to deliver these interventions in English. Thus, all subjects must be fluent in English.
7. Severe cognitive deficits that would preclude treatment with psychotherapy and/or prevent completion of study questionnaires
8. Current receipt of another form of individual psychotherapy; concurrent participation in a support group (such as Alcoholics Anonymous), couples therapy, or family therapy will be permitted
9. Currently in an abusive relationship as determined by the domestic violence questionnaire and/or PI's judgment
10. Unwilling or unable to comply with study requirements (i.e., complete forms, attend scheduled evaluations)

Exclusion Criteria (Psychiatrically Ill Children)

1. Meets criteria for mental retardation, autistic disorder, schizophrenia, or current (within prior 6 months) substance or alcohol abuse
2. Significant cognitive impairment or learning delays that would prevent completion of study questionnaires
3. Significant chronic medical illness that might explain depressive or anxiety symptoms such as sickle cell anemia, cystic fibrosis, or leukemia; children with moderate medical illnesses may be included in the study if the PI determines it is of no greater risk to the child's medical illness
4. Unwilling or unable to comply with study requirements (i.e., complete forms, attend scheduled evaluations)

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2009-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
We will compare the effects of two interventions IPT-MOMS and BSP on children outcomes: depressive symptoms (as measured by the CDI), total difficulties (as measured by the SDQ), and psychosocial functioning (as measured by the CIS) over time | Baseline, Months 3, 6, 9, 12
We will compare the two groups in depressive symptoms (as measured by the HRSD-25) and psychosocial and vocational functioning (as measured by the IIP, ISEL, and WSAS) over time. | Baseline, Months 3, 6, 9, 12

SECONDARY OUTCOMES:
We will look at major depressive episode criteria for all mothers | 3, 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Holly Swartz, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swartz HA, Cyranowski JM, Cheng Y, Zuckoff A, Brent DA, Markowitz JC, Martin S, Amole MC, Ritchey F, Frank E. Brief Psychotherapy for Maternal Depression: Impact on Mothers and Children. J Am Acad Child Adolesc Psychiatry. 2016 Jun;55(6):495-503.e2. doi: 10.1016/j.jaac.2016.04.003. Epub 2016 Apr 7. PMID 27238068